CLINICAL TRIAL: NCT06725667
Title: Ultrasound-Guided Transversalis Fascia Plane Block Versus Caudal Block for Postoperative Analgesia in Children Undergoing Inguinal Herniorrhaphy: A Randomized Controlled Non-Inferiority Trial
Brief Title: Ultrasound-Guided Transversalis Fascia Plane Block Versus Caudal Block for Postoperative Analgesia in Children Undergoing Inguinal Herniorrhaphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR935/11/24
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ultrasound; Transversalis Fascia Plane Block; Caudal Block; Postoperative Analgesia; Children; Inguinal Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis fascia plane block group (Experimental): Patients will receive transversalis fascia plane block after the induction of general anesthesia.
  Interventions: Other: Transversalis fascia plane block
- Caudal block group (Active Comparator): Patients will receive caudal block after the induction of general anesthesia.
  Interventions: Other: Caudal block

INTERVENTIONS:
Other: Transversalis fascia plane block — Patients will receive transversalis fascia plane block after the induction of general anesthesia.
  Arms: Transversalis fascia plane block group
Other: Caudal block — Patients will receive caudal block after the induction of general anesthesia.
  Arms: Caudal block group

SUMMARY:
The aim of this study is to compare ultrasound-guided transversalis fascia plane block and caudal block for postoperative analgesia in children undergoing inguinal herniorrhaphy.

DETAILED DESCRIPTION:
Surgical repair of inguinal hernia is one of the most common day-case surgeries in the pediatric population. It is associated with significant postoperative pain and discomfort.

Caudal block analgesia is a popular and reliable technique for lower abdominal surgeries and found to be safe and effective for providing intra and postoperative analgesia in pediatric patients.

transversal fascia plane block (TFPB) aims to provide analgesia for invasive procedures of the inguinal and sublingual areas by blocking the subcostal (T12), ilioinguinal (L1) and iliohypogastric (T12-L1) nerves. Several studies have reported TFPB as the analgesic method of choice for procedures involving the T12-L1 dermatome region, including iliac bone graft harvesting, cesarean section, and inguinal hernia repair

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 to 7 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for inguinal herniorrhaphy under general anesthesia (GA).

Exclusion Criteria:

* Repeated surgeries.
* Known allergic reactions to any of the study's drugs.
* Infection at the site of block needle entry.
* Bleeding diathesis.
* Neurological disorders.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-12-06 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of paracetamol administrated).

SECONDARY OUTCOMES:
Total paracetamol consumption | 24 hours postoperatively
  Each of the five items of the Face, legs, activity, cry, and consolability (FLACC) scale will be scared, ranging from 0 to 2, which will be then aggregated to obtain a total score ranging from 0 to 10. Higher scores on the scale indicated a higher level of pain intensity. If the FLACC scale exceeds three, IV paracetamol (15 mg/kg) will be given.
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Degree of pain | 24 hours postoperatively
  Degree of pain will be assessed using the Face, legs, activity, cry, and consolability (FLACC) scale. Each of the five items of the FLACC scale will be scared, ranging from 0 to 2, which will be then aggregated to obtain a total score ranging from 0 to 10. Higher scores on the scale indicated a higher level of pain intensity.
Hear rate | Every 15 min till the end of surgery (Up to 2 hours)
  Hear rate will be recorded preoperatively, before performing of block, and every 15 min till the end of surgery.
Mean arterial pressure | Every 15 min till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively, before performing of block, and every 15 min till the end of surgery.
Degree of patient's parents satisfaction | 24 hours postoperatively
  Degree of patient's parents satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication related to block such as hematoma, neurological injury, deep visceral injury, or local anesthetic toxicity will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.